CLINICAL TRIAL: NCT06163495
Title: Screen Free Time With Friends: a Cluster-randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Anders Groentved, Professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NNF20SH0062965_2
Record Dates: First submitted 2023-11-17; First posted 2023-12-11 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Time Face to Face With Friends; Screen Media Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants will engage in the Screen Free Time with Friends intervention that includes the following components:
  1. For each participating class, children and parents will be invited to two family workshops.
  2. In the beginning of 4th grade, parents will engage in a short exercise focusing on screen media use.
  3. Children will engage in school hour workshops focusing on the class culture related to screen media use and face-to-face interaction with peers.
  4. Afterschool club personal will engage in a training program consisting of three workshops aimed to increase participation rate in the afterschool club.
  5. Local stakeholders relevant to children's leisure time will engage in two workshops to develop local actions focusing on children's engagement in face-to-face interactions with peers.
  Interventions: Behavioral: Screen Free Time with Friends intervention
- Control group (No Intervention): Participants are encouraged to continue as usual.

INTERVENTIONS:
Behavioral: Screen Free Time with Friends intervention — School-based extracurricular intervention focusing on time spent with friends and screen media use
  Arms: Intervention group

SUMMARY:
The Screen Free Time with Friends study is a cluster-randomized controlled trial aiming to promote more time face-to-face with friends and reduce recreational screen media use after school and during weekends among children aged 9-11 years. The primary aim is to investigate the between group difference in change in children's time spend face-to-face with peers. Secondary aims are to investigate the between group difference in change in children's screen media use, physical activity, wellbeing, social relations, smartphone addiction, sleep and parents smartphone use and risk of smartphone addiction.

DETAILED DESCRIPTION:
During the past fifteen years, children's leisure time spent interacting with friends in person has decreased, while the time they spend engaging with digital screens has increased. These changes in behavior can potentially have adverse effects on both their physical and mental wellbeing.

This cluster-randomized controlled trial aims to evaluate an intervention aiming to increase face-to-face interaction with peers and reduce screen media use in 3rd - 4th grade-children. The study is built upon experiences gained from a recently conducted non-randomized single group feasibility trial. The feasibility trial aimed to 1) examine the feasibility of the intervention 2) examine participant recruitment and retention rates, 3) examine the feasibility of the data collection plan and completeness of the compliance and outcome assessment, and 4) obtain baseline and follow-up data on the planned full trial primary outcome.

To recruit schools and afterschool clubs for the RCT, schools will be contacted directly by a member of the research team or via the municipality. Schools and their belonging afterschool clubs are eligible if they meet the following criteria:

1. the school must have an afterschool or youth club (or similar) within walking distance,
2. the afterschool club's leader and staff must be willing to develop the club by participating in a training course.

After the baseline measurements the schools and afterschool clubs will be randomized into an intervention and control group. The Screen Free Time with Friends intervention is targeted children in 3rd to 4th grade and their families, school- and afterschool club staff, as well as stakeholders in the local community. It comprises an initial gathering for all stakeholders, family workshops held at the school, an exercise during a parent-school meeting, lectures conducted during school hours, a training program for afterschool club staff, and workshops involving local stakeholders.

A process evaluation will be conducted to monitor the implementation of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* the school must have an afterschool or youth club (or similar) within walking distance
* the afterschool club's leader and staff must be willing to develop the club by participating in a training course.

Exclusion Criteria:

* no exclusion criteria

Ages: 8 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Between group difference in change in children's time spend face-to-face with peers during leisure time at weekdays and weekenddays | Baseline and 16 months follow-up
  Children's time spent face-to-face with peers during leisure time at weekdays and weekenddays will be parent-reported at baseline and 16 months follow-up.

SECONDARY OUTCOMES:
Between group difference in change in children's time spent in afterschool club | Baseline and 16 months follow-up
  Children's time spent in an afterschool club will be parent-reported at baseline and 16 months follow-up.
Between group difference in change in children's time spent with organized activities (e.g., sport, music) during leisure time at weekdays and weekenddays | Baseline and 16 months follow-up
  Children's time spent with organized activities during leisure time at weekdays and weekenddays will be parent-reported at baseline and 16 months follow-up.
Between group difference in change in children's time spent with unorganized activities (e.g., playdates) during leisure time at weekdays and weekenddays | Baseline and 16 months follow-up
  Children's time spent with unorganized activities (e.g., playdates) during leisure time at weekdays and weekenddays will be parent-reported at baseline and 16 months follow-up.
Between group difference in change in children's time spent using screen media alone during leisure time at weekdays and weekenddays | Baseline and 16 months follow-up
  Children's time spent using screen media alone during leisure time at weekdays and weekenddays will be parent-reported at baseline and 16 months follow-up.
Between group difference in change in time in children's physical activity (any physical active behaviour) during leisure time at weekdays and weekenddays | Baseline and 16 months follow-up
  Children's physical activity (any physical active behaviour) will be assessed by Axivity AX3 triaxial accelerometers worn at the thigh using two adhesive patch 24 hours/day for seven consecutive days at baseline and 16 months follow-up.

OTHER OUTCOMES:
Between group difference in change in children's time spend face-to-face with peers during leisure time at weekdays and weekenddays | Baseline and 8 months follow-up
  Children's time spent face-to-face with peers during leisure time at weekdays and weekenddays will be parent-reported at baseline and 8 months follow-up.
Between group difference in change in children's time spend face-to-face with peers during leisure time at weekdays and weekenddays | 8 and 16 months follow-up
  Children's time spent face-to-face with peers during leisure time at weekdays and weekenddays will be parent-reported at 8 and 16 months follow-up
Between group difference in change in children's time spent in afterschool club | Baseline and 8 months follow-up
  Children's time spent in an afterschool club will be parent-reported baseline and 8 months follow-up.
Between group difference in change in children's time spent in afterschool club | 8 and 16 months follow-up
  Children's time spent in an afterschool club will be parent-reported at 8 and 16 months follow-up.
Between group difference in change in children's time spent with organized activities (e.g., sport, music) during leisure time at weekdays and weekenddays | Baseline and 8 months follow-up
  Children's time spent with organized activities during leisure time at weekdays and weekenddays will be parent-reported at baseline and 8 months follow-up.
Between group difference in change in children's time spent with organized activities (e.g., sport, music) during leisure time at weekdays and weekenddays | 8 and 16 months follow-up
  Children's time spent with organized activities during leisure time at weekdays and weekenddays will be parent-reported at 8 and 16 months follow-up.
Between group difference in change in children's time spent with unorganized activities (e.g., playdates) during leisure time at weekdays and weekenddays | Baseline and 8 months follow-up
  Children's time spent with unorganized activities (e.g., playdates) during leisure time at weekdays and weekenddays will be parent-reported at baseline and 8 months follow-up.
Between group difference in change in children's time spent with unorganized activities (e.g., playdates) during leisure time at weekdays and weekenddays | 8 and 16 months follow-up
  Children's time spent with unorganized activities (e.g., playdates) during leisure time at weekdays and weekenddays will be parent-reported 8 and 16 months follow-up.
Between group difference in change in children's time spent using screen media alone during leisure time at weekdays and weekenddays | Baseline and 8 months follow-up
  Children's time spent using screen media alone during leisure time at weekdays and weekenddays will be parent-reported at baseline and 8 months follow-up.
Between group difference in change in children's time spent using screen media alone during leisure time at weekdays and weekenddays | 8 and 16 months follow-up
  Children's time spent using screen media alone during leisure time at weekdays and weekenddays will be parent-reported at 8 and 16 months follow-up.
Between group difference in change in children's smartphone time at weekdays and weekenddays | Baseline and 16 months follow-up
  Children's smartphone time at weekdays and weekenddays will be assessed objectively continuously during the intervention by an application installed on the participants devices and extrapolated from their smartphone.
Between group difference in change in children's smartphone time at weekdays and weekenddays | Baseline and 8 months follow-up
  Children's smartphone time at weekdays and weekenddays will be assessed objectively continuously during the intervention by an application installed on the participants devices and extrapolated from their smartphone.
Between group difference in change in children's smartphone time at weekdays and weekenddays | 8 and 16 months follow-up
  Children's smartphone time at weekdays and weekenddays will be assessed objectively continuously during the intervention by an application installed on the participants devices and extrapolated from their smartphone.
Between group difference in change in children's total screen time at weekdays and weekenddays | Baseline and 16 months follow-up
  Children's total screen time at weekdays and weekenddays will be parent-reported at baseline and follow-up. Also, children's screen use before bedtime will be parent-reported at baseline and 16 months follow-up.
Between group difference in change in children's time in moderate to vigorous physical activity (MVPA) during leisure time at weekdays and weekenddays | Baseline and 16 months follow-up
  Children's moderate to vigorous physical activity (MVPA) during leisure time at weekdays and weekenddays will be assessed by Axivity AX3 triaxial accelerometers worn at the thigh using two adhesive patch 24 hours/day for seven consecutive days at baseline and 16 months follow-up.
Between group difference in change in children's wellbeing | Baseline and 16 months follow-up
  The wellbeing of the children will be measured using the Danish version of the Strengths and Difficulties Questionnaire (SDQ) for teachers at baseline and 18 months follow-up. In addition, children's wellbeing will be self-reported using a child questionnaire including the Cantril's scale rating from 10 (the best possible life) to 0 (the worst possible life). Furthermore, children will answer a question about loneliness answered on a four-point Likert scale.
Between group difference in change in children's social relations | Baseline and 16 months follow-up
  Social network analysis will be employed to examine the children's social relationships within the class.
Between group difference in change in school class cohesion | Baseline and 16 months follow-up
  Children will answer questions related to school class cohesion (e.g., sense of belonging) at baseline and 16 months follow-up.
Between group difference in change in children's screen media addiction | Baseline and 16 months follow-up
  Children's screen media addiction will be parent-reported using the Problematic Media Use Measure Short Form (PMUM-SF).
Between group difference in change in children's sleep | Baseline and 16 months follow-up
  Children's sleep will be assessed seven consecutive days at baseline and 16 months follow-up using the Axivity AX3 triaxial accelerometers. The objective measures of sleep duration will be supplemented by few questions about sleep in the parental questionnaire.
Between group difference in change in parent's smartphone use at weekdays and weekenddays | Baseline 16 months follow-up
  Parent's smartphone time at weekdays and weekenddays will be assessed objectively continuously during the intervention by an application installed on the participants devices.
Between group difference in change in parent's smartphone use at weekdays and weekenddays | Baseline and 8 months follow-up
  Parent's smartphone time at weekdays and weekenddays will be assessed objectively continuously during the intervention by an application installed on the participants devices.
Between group difference in change in parent's smartphone use at weekdays and weekenddays | 8 and 16 months follow-up
  Parent's smartphone time at weekdays and weekenddays will be assessed objectively continuously during the intervention by an application installed on the participants devices.
Between group difference in change in parent's smartphone addiction | Baseline and 16 months follow-up
  The smartphone addiction scale - short version (SAS-SV) consisting of 10 items rated on a 6-point Likert scale (strongly disagree to strongly agree) will be used to assess the level of risk of smartphone addiction among parents.
Between group difference in change in children's time spent face-to-face with family during leisure time at weekdays and weekenddays | Baseline and 16 months follow-up
  Children's time spent face-to-face with family during leisure time at weekdays and weekenddays will be self-reported and parent-reported at baseline and 16 months follow-up.
Between group difference in change in children's online communication | Baseline and 16 months follow-up
  Children will answer questions related to online communication such as amount and experiences at baseline and 16 months follow-up.
Between group difference in change in parent's awareness of and attitude towards screen media use | Baseline and 16 months follow-up
  Parents will answer questions about their awareness and attitude towards screen media use at baseline and 16 months follow-up.
Between groups difference in change in dialogue in the family | Baseline and 16 months follow-up
  At baseline and 16 months follow-up, parents will answer questions about whether and how parents and children discuss/talk about aspects related to screen media use.
Between group difference in change in family screen media rules | Baseline and 16 months follow-up
  At baseline and 16 months follow-up, parents will answer questions about family screen media rules, which also encompass the children's satisfaction with these (potential) rules.
Between group difference in change in conflicts rooted in screen media use (in the family) | Baseline and 16 months follow-up
  At baseline and 16 months follow-up, parents will answer questions about the frequency of conflicts rooted in screen media use in the family.
Between group difference in change in parent's awareness and attitude towards children's leisure time activities | Baseline and 16 months follow-up
  At baseline and 16 months follow-up, parents will answer questions about awareness and attitude towards children's leisure time activities including the afterschool program.
Between group difference in change in dialogue among parents (in a school class) | Baseline and 16 months follow-up
  At baseline and 16 months follow-up, parents will answer questions about whether parents in the school class discuss aspects related to screen media use, the afterschool program, or leisure time activities.
Change in perceived network and motivation among local stakeholders | Baseline and 16 months follow-up
  At baseline and 16 months follow-up, local stakeholders in the intervention group will answer questions related to their perceived social network and motivation for improving children's opportunities to spend time face-to-face with peers in the local community.
Amount and type of actions initiated by local stakeholders | 8 and 16 months follow-up
  At 8 and 16 months follow-up local stakeholders in the intervention group will answer questions about the amount and type of local actions initiated as a result of the local workshops.
Amount and type of actions initiated by the afterschool staff | 8 and 16 months follow-up
  At 8 and 16 months follow-up the afterschool staff in the intervention group will answer questions about the amount and type of actions initiated as a result of the training program.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Grøntved, PhD, Principal Investigator — Department of Sports Science and Clinical Biomechanics, University of Southern Denmark
Locations (18):
- Denmark (18):
  - Bregnbjergskolen, Vojens, Haderslev
  - Spjald skole, Spjald, Ringkøbing
  - Auraskolen, Bryndum skole, Esbjerg
  - Auraskolen, Hjerting skole, Esbjerg
  - Auraskolen, Sønderrisskolen, Esbjerg
  - Mørkhøj skole, Gladsaxe
  - Holmegaardskolen, Næstved
  - Vesterlandsskolen, Næstved
  - Kroggårdskolen, Odense
  - Næsby skole, Odense
  - Skt. Klemensskolen, Odense
  - Søhusskolen, Odense
  - Kildeskolen, Ringsted
  - Nordbakkeskolen, Ringsted
  - Hvinningdalskolen, Silkeborg
  - Resenbro skole, Silkeborg
  - Sorring Skole, Silkeborg
  - Skolen i Skjern, Skjern

IPD SHARING:
Plan to Share IPD: No